CLINICAL TRIAL: NCT07020897
Title: Short-term and Intermediate-term Effects of Self-applied Joint Mobilization Versus Clinician-applied Joint Mobilization in Addition to Exercise in Patients With Knee Osteoarthritis: A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Texas Health Resources (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-FY2025-156
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee flexion contracture; Knee osteoarthritis; Joint mobilization; Physical therapy; Hip abductor strength
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinician-administered joint mobilization (Active Comparator): In-clinic exercise-based physical therapy, home exercise program, and clinician-administered joint mobilization.
  Interventions: Other: Clinician-administered joint mobilization; Other: Exercise-based physical therapy
- Self-administered joint mobilization (Experimental): In-clinic exercise-based physical therapy, home exercise program, and self-administered joint mobilization.
  Interventions: Other: Self-administered joint mobilization; Other: Exercise-based physical therapy

INTERVENTIONS:
Other: Clinician-administered joint mobilization — Tibiofemoral arthrokinematic extension joint mobilization and multidirectional patellofemoral mobilization applied by a physical therapist.
  Arms: Clinician-administered joint mobilization
Other: Self-administered joint mobilization — Tibiofemoral arthrokinematic extension joint mobilization and multidirectional patellofemoral mobilization applied by the research participant.
  Arms: Self-administered joint mobilization
Other: Exercise-based physical therapy — In-clinic exercise-based physical therapy supervised by a physical therapist, with home exercises to be performed on days without a clinical visit.

SUMMARY:
The goal of this clinical trial is to learn if a combination of patient self-administered joint mobilization and exercise works to treat knee osteoarthritis in adults. The main questions it aims to answer are:

* Does self-administered joint mobilization improve the ability to perform regular daily activities?
* Does self-administered joint mobilization improve knee motion?
* Does self-administered joint mobilization improve hip strength?

Researchers will compare the program of self-administered joint mobilization to a joint mobilization administered by a physical therapist.

Participants will:

* Attend 8-12 physical therapy clinic visits over 6 - 8 weeks
* Perform home exercises
* Visit the clinic 6 months later for a brief check-up

DETAILED DESCRIPTION:
This study will take place in the Outpatient Rehabilitation Clinic at Texas Health Resources (THR) in Plano, or in the Texas Health Sports Medicine Clinic in Allen.

Participants in this study will be asked to complete the same intake forms and questionnaires as any other physical therapy patient being seen for knee pain at all of the THR physical therapy clinics. These will include questions about health history, learning style, living situation, and goals for physical therapy treatment. One investigator will perform a physical therapy evaluation, including joint motion, muscle strength, and flexibility measurements, as well as functional testing.

For this study, we will measure one knee motion and one hip strength item and ask participants to complete a knee- specific questionnaire 3 times: on the initial evaluation visit, during the last visit of physical therapy, and during a 6-month follow-up visit.

After the initial evaluation visit, we will assign each participant into one of the two treatment groups, self-joint mobilization or joint mobilization performed by a physical therapist. Participants will be asked to attend 7 - 11 physical therapy treatment visits over 7-8 weeks for strength training exercises, flexibility exercises, joint mobilization, and a home exercise program. Each physical therapy visit, including the initial evaluation visit will last 45 minutes. Participants will be asked to track compliance with a home program and attend a follow-up appointment about 6 months after the initial evaluation. This follow-up visit will last about 30 minutes.

All appointments, except for the 6-month follow-up, will be structured and carried out as they would for any other patient receiving physical therapy for knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Meets National Institute for Health and care Excellence (NICE) criteria for knee osteoarthritis:
* Age 45 years or older
* Movement-related knee pain
* No morning stiffness or morning stiffness < 30 minutes
* Knee flexion contracture (kFC) at least 1cm, measured by heel-height
* Fluency in verbal and written English for completion of outcome measure and screening, and to take directions.
* Able to attend all study-related appointments

Exclusion Criteria:

* Assistive device required for ambulation
* Systemic disease affecting joint function (diabetes, rheumatological disorders, etc)
* Previous lower extremity joint replacement
* Lower quarter surgery, injection, or therapy in the past year
* Other functionally-limiting physical impairment of the lower quarter
* Spine or lower extremity compensation claim (work, accident, etc)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Baseline (enrollment), 6-8 weeks (end of physical therapy sessions), 6 months
  The WOMAC is a self-administered questionnaire assessing pain, stiffness, and physical function in patients with knee osteoarthritis.

SECONDARY OUTCOMES:
Hip abductor strength | Baseline (enrollment), 6-8 weeks (end of physical therapy sessions), 6 months
  Hip abductor strength measured by hand-held dynamometer
Passive knee extension range of motion | Baseline (enrollment), 6-8 weeks (end of in-clinic physical therapy), 6 months
  Passive knee extension range of motion will be measured in supine with traditional goniometry and in prone with a heel-height measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Guy L Terry, MPT, PhD(c), Principal Investigator — Texas Woman's University
Locations (2):
- United States (2):
  - Texas Health Resources Sports Medicine Allen, Allen, Texas
  - Texas Health Resources Plano Presbyterian Outpatient Rehabilitation, Plano, Texas

IPD SHARING:
Plan to Share IPD: No
Sharing IPD raises ethical concerns about participant privacy and the potential for misuse of sensitivity data. Data protection laws and regulations can restrict the sharing of personal data, even for research purposes.